CLINICAL TRIAL: NCT01314833
Title: Adjuvant 6 Cycles of Docetaxel and Cyclophosphamide or 3 Cycles of Cyclophosphamide/Epirubicin/Fluorouracil Followed by 3 Cycles of Docetaxel Versus 4 Cycles of Epirubicin and Cyclophosphamide Followed by Weekly Paclitaxel in HER2-negative Operable Breast Cancer
Brief Title: Minus Anthracycline or Short-Term Versus Epirubicin and Cyclophosphamide Followed by Paclitaxel Regimen for Adjuvant Breast Cancer Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Chinese Anti-Cancer Association (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MASTER
Record Dates: First submitted 2011-03-09; First posted 2011-03-15 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Primary Breast Cancer
Keywords: Luminal A; Luminal B; TNBC; DFS; DDFS; OS
MeSH Terms: interventions — CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TC*6 (Experimental): 6 cycles of (Docetaxel 75mg/m2 ivgtt d1+ Cyclophosphamide 600 mg/m2 iv d1, 21 days per cycle) .
  Interventions: Drug: Docetaxel Cyclophosphamide
- CEF*3-T*3 (Experimental): 3 cycles of CEF (Epirubicin 100 mg/m2 ivgtt d1+Cyclophosphamide 500 mg/m2 iv d1+ 5-fluorouracil 500 mg/m2 iv d1, 21 days per cycle) followed by 3 cycles of Docetaxel (Docetaxel 100mg/m2, ivgtt d1, 21 days per cycle)
  Interventions: Drug: Cyclophosphamide Fluorouracil Epirubicin Docetaxel
- EC*4-wP*12 (Experimental): 4 cycles of EC (Epirubicin 90 mg/m2 ivgtt d1+Cyclophosphamide 600 mg/m2 iv d1, 21 days per cycle) followed by 4 cycles of Paclitaxel (Paclitaxel 80mg/m2, ivgtt d1,8,15, 21days per cycle)
  Interventions: Drug: Epirubicin Cyclophosphamide Paclitaxel

INTERVENTIONS:
Drug: Docetaxel Cyclophosphamide — Docetaxel 75 mg/m² D1 Cyclophosphamide 600 mg/m² D1
  1 cycle = 21 days
  TC*6
  Arms: TC*6
Drug: Cyclophosphamide Fluorouracil Epirubicin Docetaxel — 1st -3rd Cycle: Fluorouracil 500 mg/m² D1 Epirubicin 100 mg/m² D1 Cyclophosphamide 500 mg/m² D1
  1 cycle = 21 days
  4th-6th Cycle: Docetaxel 100mg/m² D1
  1 cycle = 21 days CEF*3-T*3
  Arms: CEF*3-T*3
Drug: Epirubicin Cyclophosphamide Paclitaxel — 1st-4th Cycle: Epirubicin 90 mg/m² D1 Cyclophosphamide 600 mg/m² D1
  1 cycle = 21 days
  5th-8th Cycle: Paclitaxel 80mg/m² D1, 8, 15
  1 cycle = 21 days EC*4-P*4
  Arms: EC*4-wP*12

SUMMARY:
We aimed to evaluate the noninferiority of short-term anthracycline-free chemotherapy (TC, six cycles of docetaxel and cyclophosphamide) or short-term anthracycline-based chemotherapy (CEF-T, three cycles of cyclophosphamide/epirubicin/fluorouracil followed by three cycles of docetaxel) to a standard anthracycline/taxane-containing chemotherapy (EC-P, epirubicin, and cyclophosphamide for four cycles followed by paclitaxel for twelve weeks) in HER2-negative operable breast cancer.

DETAILED DESCRIPTION:
It was initiated as an adjuvant chemotherapy trial to test noninferiority of an anthracycline-free short-term regimen (T75C600 x 6 [TC] once every 3 weeks) or a short-term regimen (C500E100F500 x 3 once every 3 weeks followed by T100 x 3 every 3 weeks [CEF-T]) compared with a standard long-term anthracycline-containing regimen (E90C600 x 4 once every 3 weeks followed by P80 x 12 once every week [EC-P]) in HER2-negative breast cancer. Patients were randomly assigned (1:1:1) to each arm after completing the surgical excision of the primary tumor.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age at diagnosis 18 - 75 years
* Histological confirmed unilateral primary invasive carcinoma of the breast
* Adequate surgical treatment with complete resection of the tumor (R0) and resection of > or = 10 axillary nodes or SLN in clinically N0 patients
* Node positive disease or node-negative disease with at least one other risk factor (tumor size > or = 2 cm, grade > or = II)
* HER2-negative disease
* No evidence for distant metastasis (M0) after conventional staging
* Performance Status ECOG < or = 1
* The patient must be accessible for treatment and follow-up
* LVEF> 50%
* Negative pregnancy test (urine or serum) within 7 days prior to randomization in premenopausal patients
* Leucocytes > or = 4 x 10^9/L
* platelets > or = 100 x 10^9/L
* haemoglobin > or = 9 g/dL
* total bilirubin < or = 1.5 UNL
* ASAT (SGOT) and ALAT (SGPT) < or = 2.5 UNL
* creatinine < 175 mmol/L (2 mg/dL)

Exclusion Criteria:

1. Has received neoadjuvant therapy (include chemotherapy, targeted therapy, radiotherapy or endocrine therapy）;
2. Has bilateral breast cancer;
3. Has the previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ.
4. Has metastatic (Stage 4) breast cancer;
5. Has any >T4 lesion (UICC1987) (with skin involvement, mass adhesion and fixation, and inflammatory breast cancer);
6. Is pregnant, is breastfeeding women, or women of childbearing age who cannot practice effective contraceptives;
7. Patients participating in other clinical trials at the same time;
8. Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmgh, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
9. Has known allergy to taxane and excipients;
10. Has severe or uncontrolled infection.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1570 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Disease-Free Survival | 5 years
  Defined as the time from randomization to occurrence of a new event including local recurrence, regional relapse, distant metastasis, contralateral primary breast cancer, second non-breast invasive cancer (excluding non-melanoma skin cancers), or death from any cause.

SECONDARY OUTCOMES:
Distant Disease-Free Survival | 5 years
  Defined as the time from randomization to the earliest recurrence outside of the ipsilateral locoregional region or to death from any cause, whenever a death occurred before distant recurrence
Overall Survival | 5 years
  defined as the time from randomization to death from any cause
Adverse Events | through chemotherapy completion, an average of 6 months
  Number of Participants with Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones S, Holmes FA, O'Shaughnessy J, Blum JL, Vukelja SJ, McIntyre KJ, Pippen JE, Bordelon JH, Kirby RL, Sandbach J, Hyman WJ, Richards DA, Mennel RG, Boehm KA, Meyer WG, Asmar L, Mackey D, Riedel S, Muss H, Savin MA. Docetaxel With Cyclophosphamide Is Associated With an Overall Survival Benefit Compared With Doxorubicin and Cyclophosphamide: 7-Year Follow-Up of US Oncology Research Trial 9735. J Clin Oncol. 2009 Mar 10;27(8):1177-83. doi: 10.1200/JCO.2008.18.4028. Epub 2009 Feb 9. PMID 19204201